CLINICAL TRIAL: NCT03156855
Title: Comparison of the Efficacy of Sequential Therapy and Bismuth Quadruple Therapy in the First Line and Second Line Therapy for Helicobacter Pylori Infection- A Multi-center Randomized Trial
Brief Title: Sequential Therapy Versus Quadruple Therapy in H. Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: E-DA Hospital (Other); National Taiwan University Hospital Hsin-Chu Branch (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Kaohsiung Medical University (Other); Chiayi Christian Hospital (Other); Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201506129MINC
Record Dates: First submitted 2015-09-30; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Helicobacter
Keywords: efficacy; safety; H. pylori eradication
MeSH Terms: interventions — ribosomal protein S14; Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sequential therapy for 14 days (S14) (Experimental): 14 day sequential therapy
  Interventions: Drug: 14-day sequential therapy
- bismuth quadruple therapy (Q10) (Active Comparator): Bismuth quadruple therapy
  Interventions: Drug: Bismuth quadruple therapy

INTERVENTIONS:
Drug: 14-day sequential therapy — D1-D7: (esomeprazole 40mg qid + amoxicillin 500mg qid) for 7 days D8-D14: (esomeprazole 40mg qid + clarithromycin 500mg bid + metronidazole 500mg bid) for another 7 days
  Other Names: S14
  Arms: sequential therapy for 14 days (S14)
Drug: Bismuth quadruple therapy — D1-D10: (esomeprazole 40mg bid + dibismuth trioxide 120mg qid + metronidazole 500mg tid + tetracycline 500mg qid) for 10 days
  Other Names: Q10
  Arms: bismuth quadruple therapy (Q10)

SUMMARY:
The investigators aimed to

1. compare the eradication rates and long term re-infection rates of sequential therapy for 14 days versus bismuth quadruple therapy for 10 days in the first line and second line treatment
2. assess the impact of antibiotic resistance and CYP2C19 polymorphism on the eradication rate of these regimens
3. assess the impact of these eradication regimens on the antibiotic resistance and microbiota of the gut flora
4. assess the impact of eradication therapy on the metabolic factors

DETAILED DESCRIPTION:
Helicobacter pylori infection has been shown to be associated with the development of gastric cancer and peptic ulcer diseases. Eradication of H. pylori infection reduces the risk of gastric cancer and recurrence of peptic ulcer disease. However, the eradication rate of clarithromycin-based triple therapy has been declining in recent years, probably related to the increasing resistant rate to clarithromycin. Sequential therapy for 10 days has been shown to be more effective than triple therapy for 7 and 10 days. The investigators further demonstrated that sequential therapy given for 14 days was superior to triple therapy given for 14 days. Recently, the investigators also found that bismuth quadruple therapy given for 10 days appeared to be more effective than triple therapy given for 14 days in the first line therapy. However, whether sequential therapy given for 14 days is more effective than bismuth quadruple therapy or triple therapy for 14 days remains unknown.

ELIGIBILITY:
Inclusion Criteria:

1. H. pylori infected patients naïve to eradication therapies will be eligible in this study.

Exclusion Criteria:

1. children and teenagers aged less than 20 years,
2. history of gastrectomy,
3. gastric malignancy, including adenocarcinoma and lymphoma,
4. previous allergic reaction to antibiotics (bismuth, amoxicillin, metronidazole, clarithromycin, tetracycline) and PPI (esomeprazole),
5. contraindication to treatment drugs,
6. pregnant or lactating women,
7. severe concurrent disease,
8. concomitant use of clopidogrel, or (9) Unwilling to accept random assignment of subjects

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate: determined by urea breath test (13C-UBT, according to ITT analysis) | 6 weeks
  No eradicated divided by total cases by intention to treat analysis. 13C-UBT will be used to determine the H. pylori status at least 6 weeks after completion of treatment. A delta value of > 4 units will be defined as positive for H. pylori infection as our previous studies.

SECONDARY OUTCOMES:
adverse effect: occurrence of any adverse effect during the treatment | 2 weeks
  adverse effects related to treatment by per protocol analysis. The patients will be informed of the common side effects from the studied drugs prior to therapy. They will also be asked to record these symptoms during treatment. A standardized interview at the outpatient clinic at the end of treatment will be arranged. The adverse events and compliance will be assessed by the research staffs with pre-defined case report form.
changes of antibiotic resistance | 2 weeks, 8 weeks, 1 year
  changes of antibiotic resistance of E. coli by per protocol analysis

OTHER OUTCOMES:
changes of gut microbiota | 2 weeks, 8 weeks, 1 year
  changes of gut microbiota before and after HP eradication by per protocol analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, PhD, Study Director — National Taiwan University Hospital
Locations (7):
- Taiwan (7):
  - Chiayi Christian Hospital, Chiayi City
  - National Taiwan University Hospital, Hsinchu Branch, Hsinchu
  - E-DA University Hospital, Kaohsiung City
  - Jyh-Ming Liou, Taipei
  - Taipei Veteran General Hospital, Taipei
  - Mackay Memorial Hospital, Taitung branch, Taitung
  - National Taiwan University Hospital, Yun-Lin Branch, Yunlin County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liou JM, Chen CC, Fang YJ, Chen PY, Chang CY, Chou CK, Chen MJ, Tseng CH, Lee JY, Yang TH, Chiu MC, Yu JJ, Kuo CC, Luo JC, Hsu WF, Hu WH, Tsai MH, Lin JT, Shun CT, Twu G, Lee YC, Bair MJ, Wu MS; Members of the Taiwan Gastrointestinal Disease and Helicobacter Consortium. 14 day sequential therapy versus 10 day bismuth quadruple therapy containing high-dose esomeprazole in the first-line and second-line treatment of Helicobacter pylori: a multicentre, non-inferiority, randomized trial. J Antimicrob Chemother. 2018 Sep 1;73(9):2510-2518. doi: 10.1093/jac/dky183. PMID 29846605